CLINICAL TRIAL: NCT05507346
Title: A Multi-center Randomized Control Cross-over Study to Evaluate the Effectiveness of a Novel Portable Non-Pneumatic Active Compression Device vs. an Advanced Pneumatic Compression Device for Treating Lower Extremity Lymphedema (TEAYS)
Brief Title: A Clinical Study to Evaluate the Effectiveness of a Novel Portable Non-Pneumatic Active Compression Device vs. an Advanced Pneumatic Compression Device for Treating Lower Extremity Lymphedema
Acronym: TEAYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koya Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KCT 009 (TEAYS)
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2024-03

CONDITIONS: Lymphedema; Lymphedema of Leg; Chronic Venous Insufficiency; Venous Insufficiency; Lymphedema, Lower Limb
MeSH Terms: conditions — Lymphedema; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dayspring, Non-Pneumatic Active Compression Device (NPCD) (Experimental): The Dayspring, an Non-Pneumatic Active Compression Device (NPCD) Active Wearable Compression Device is an FDA cleared calibrated active gradient pressure compression garment that is segmental and programmable and applies controlled sequential pressure from the distal to proximal-end of the limb in a cyclic manner.
  Interventions: Device: Cross over Device (PCD or Dayspring - alternate to first group)
- Advanced Pneumatic Compression Device (APCD) (Active Comparator): A commercially available advanced pneumatic compression device that is FDA-cleared for the same indication for use as the Dayspring Wearable Compression Device.
  Interventions: Device: Cross over Device (PCD or Dayspring - alternate to first group)

INTERVENTIONS:
Device: Cross over Device (PCD or Dayspring - alternate to first group) — Cross over after three month of use and a month of washout period

SUMMARY:
To evaluate the Koya wearable device - a Novel Portable Non-Pneumatic Active Compression Device (NPCD) in contrast to an advanced pneumatic compression device (APCD)

DETAILED DESCRIPTION:
A Multi-center Randomized Control Single Cross-over Study to Evaluate the Safety and Effectiveness of Dayspring, a Novel Portable Non-Pneumatic Active Compression Device (NPCD) vs. an Advanced Pneumatic Compression Device (APCD) for Treating Lower Extremity Lymphedema. To evaluate the Dayspring, a Novel Portable Non-Pneumatic Active Compression Device (NPCD) in contrast to an advanced pneumatic compression device (APCD) in a multi-centered setting to evaluate volume, quality of life, safety, adherence, and preference.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Capable and willing to sign the informed consent and deemed capable of following the study protocol
* Subjects must have a diagnosis of primary or secondary unilateral or bilateral lower extremity edema or lower extremity phlebolymphedema from chronic venous insufficiency

Exclusion Criteria:

* Individuals with a history or presence of a systemic disorder or condition that could place the subject at increased risk from sequential compression therapy
* Inability or unwillingness to participate in all aspects of study protocol and/or inability to provide informed consent
* Subjects with exam results that would prevent safe and effective use of the study device (cellulitis, open-wounds, healing-wounds, etc.)
* Subjects must not have any diagnosed cognitive or physical impairment that would interfere with use of the device
* Individuals who present with Ankle-brachial Index (ABI) screening score < 0.8 and > 1.30, indicating the possibility of Peripheral Arterial disease (PAD)
* Diagnosis of lipedema
* Diagnosis of active or recurrent cancer (< 3 months since completion of chemotherapy, radiation therapy or primary surgery for the cancer)
* Diagnosis of acute infection (in the last four weeks)
* Diagnosis of acute thrombophlebitis (in last 6 months)
* Diagnosis of pulmonary embolism or deep vein thrombosis within the previous 6 months
* Diagnosis of pulmonary edema
* Diagnosis of congestive heart failure (uncontrolled/uncompensated)
* Diagnosis of chronic kidney disease with acute renal failure
* Diagnosis of epilepsy
* Subjects with poorly controlled asthma
* Any condition where increased venous and lymphatic return is undesirable
* Women who are pregnant, planning a pregnancy or nursing at study entry
* Participation in any clinical trial of an investigational substance or device during the past 30 days

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Limb volume reduction or maintenance | 3 months
  Limb volume measurement is performed by using a calibrated tape measure to measure circumference from the ankle at 4cm increments to the waist region. Measurements to be taken for both lowerr extremities. Volume is calculated based on cylindrical segment analysis. The outcome measure is assessed as a difference or change from baseline to month 3
LYMQOL | 3 months
  The Lymphedema Quality of Life Questionnaire (LYMQOL), a validated disease-specific QoL tool, is also administered at baseline and month 3. Overall QoL is scored on a single item by the patient on a scale of 1-10. The outcome measure is assessed as a difference or change from baseline LYMQOL at day zero and month 3
Therapy adherence tracking | 3 months
  A table will be provided to patient to document days of use with the device to track adherence

SECONDARY OUTCOMES:
Safety/AEs | 3 months
  As assessed by reported adverse events
Patient survey on preference | 3 months
  A study survey administered at the end of the study to measure patient preference between the two devices

CONTACTS AND LOCATIONS:
Locations (1):
- Stanley G Rockson, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No